CLINICAL TRIAL: NCT03439241
Title: Assessment of the Performance of a New Ostomy Device in Sub-jects Having an Ileostomy
Brief Title: Assessment of the Performance of a New Ostomy Device in Subjects Having an Ileostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CP278
Record Dates: First submitted 2018-02-12; First posted 2018-02-20 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Ileostomy - Stoma

STUDY DESIGN:
Intervention Model Description: The trial starts with a baseline period. After 4 baseplate changes the subjects is randomised into two arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Silent arm (Experimental): The participants test the new Coloplast ostomy device use the product as they usually would.
  Interventions: Device: Coloplast ostomy device
- Active arm (Experimental): The participants test the tnew Coloplast ostomy device and are guided by the measuring device
  Interventions: Device: Coloplast ostomy device

INTERVENTIONS:
Device: Coloplast ostomy device — the test product is a newly developed Coloplast ostomy device

SUMMARY:
The purpose was to investigate the performance of a new ostomy device measured with a measuring device.

ELIGIBILITY:
Inclusion Criteria:

1. Have given written informed consent and in DK: signed a letter of authority
2. Be at least 18 years of age and have full legal capacity
3. Have had their ileostomy for at least 3 months
4. Can use a product with max cut size 45 mm
5. Self-reported problems with leakage (3 x within 14 days)
6. Be willing and suitable (determined by the investigator representative) to use the test product without using a paste/mouldable ring during the test period
7. Must be able to use custom cut product
8. Minimum change of product every third day
9. Get a negative result of a pregnancy test for women of childbearing age (only DK)

Exclusion Criteria:

1. Are currently receiving or have within the past 2 months received radio-and/or chemotherapy (low doses chemotherapy is allowed for other indications than cancer, e.g. below 15 mg methotrexate for rheumatoid arthritis)
2. Are currently receiving or have within the past month received topical steroid treatment in the peristomal skin area, e.g. lotion or spray. Systemic steroid treatment (e.g. injection, or tablet) are allowed.
3. Are pregnant or breastfeeding
4. Are participating in other interventional clinical investigations or have previously participated in this investigation Exception: Participation in other Coloplast in-house clinical investigations is accepted under the circumstances that the subject has paused the activities in the investigation and are otherwise complying with the inclusion and exclusion criteria of this (CP278) protocol.
5. Are currently suffering from peristomal skin problems i.e. bleeding and/or broken skin (assessed by the investigator)
6. Have known hypersensitivity towards any of the products used in the investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-04-16 (Actual); Study Completion 2018-04-16 (Actual)

PRIMARY OUTCOMES:
wear time (hours) | 14 days
  Wear time is recorded at each baseplate change

CONTACTS AND LOCATIONS:
Overall Officials: Birte P Jakobsen, MD, Principal Investigator — Medical Director
Locations (1):
- Coloplast A/S, Humlebæk, Denmark